CLINICAL TRIAL: NCT06201468
Title: SCAPULAR MOBILIZATION VERSUS SCAPULAR PROPRIOCEPTIVE NEURO MUSCULAR FACILITATION ON FROZEN SHOUDER
Brief Title: Frozen Shoulder (Scapular Mobilization Versus Scapular PNF)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud El morsy, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Frozen shoulder
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Frozen Shoulder; Scapular Mobilization; Scapular Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Two treatment groups will receive interventions as follows:
  Group A (n = 21): will receive scapular mobilization combined with mobilization with movement (MWM) and capsular stretch for 4 weeks.
  Group B (n = 21): will receive scapular proprioceptive neuromuscular facilitation combined with (MWM) and capsular stretch for 4 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple-blinded clinical randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Group A (n = 21): will receive scapular mobilization combined with mobilization with movement (MWM) and capsular stretch for 4 weeks.
  Mulligan Mobilization with Movement for peripheral joints combines sustained manual application of 'gliding' force to a joint, with the aim of repositioning the positional faults with concurrent physiological motion of the joint, either performed actively by the subject or passively by the therapist
  Interventions: Other: Group A SCAPULAR MOBILIZATION
- group B (Experimental): Group B (n = 21): will receive scapular proprioceptive neuromuscular facilitation combined with (MWM) and capsular stretch for 4 weeks.
  Scapular PNF incorporates functional or diagonal patterns (anterior elevation - posterior depression and posterior elevation - anterior depression) for performing the exercises and can be used to stretch or strengthen the muscles selectively. These techniques help the muscles to relearn the normal timing of recruitment and the amount of activation to sustain the balance between different groups of muscles
  Interventions: Other: Group A SCAPULAR MOBILIZATION

INTERVENTIONS:
Other: Group A SCAPULAR MOBILIZATION — Two treatment groups will receive interventions as follows:
  Group A (n = 21): will receive scapular mobilization combined with mobilization with movement (MWM) and capsular stretch for 4 weeks.
  Group B (n = 21): will receive scapular proprioceptive neuromuscular facilitation combined with (MWM) and capsular stretch for 4 weeks.
  Other Names: GROUP B SCAPULAR PNF

SUMMARY:
This study will be conducted to examine and compare the effects of SM versus SPNF on shoulder pain, ROM and functional disabilities in patients with frozen shoulder.

DETAILED DESCRIPTION:
This study will be conducted to examine and compare the effects of SM versus SPNF on shoulder pain, ROM and functional disabilities in patients with frozen shoulder.

ELIGIBILITY:
Inclusion Criteria:

- All the patients refferd from orthopaedic surgeon with diagnosis of adhesive capsulitis. Patients will be included in this study if they fulfil the following criteria

1. Case diagnosed with adhesive capsulitis, both primary and secondary.
2. Both males and females of the age group 40 to 60 years.
3. Limited active and passive movement of the shoulder joint movements, as well as difficulties with ADLs.

4- The onset of symptoms between 3 to 12 months. 5. Unilateral adhesive capsulitis.

Exclusion Criteria:

* 1. History of shoulder surgery or manipulation under anaesthesia, local corticosteroid injection administration to the affected shoulder within the last 6 months, 2. Neurological deficit affecting the shoulder function during daily activities, 3. Pathology of the shoulder joint other than adhesive capsulitis including rotator cuff tear, tendonitis at the shoulder and neck region, malignancies, history of trauma or accidental injuries of the upper limb.

  4- Other pathological conditions including, a history of stroke, history of mastectomy and coronary artery bypass grafting (CABG).

  5. Rheumatoid arthritis, osteoporosis, or disorders of the cervical spine, elbow, wrist or hand.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder disability | 4 weeks
  Shoulder Pain and Disability Index (SPADI)
  The translated version of SPADI in the Arabic language showed excellent internal consistency and test-retest reliability. Validity was shown by substantial correlations between SPADI and Quick DASH, NRS, and active shoulder ROM. The Arabic SPADI is recommended for the evaluation of patients with shoulder dysfunction
Shoulder range of motion | 4 weeks
  A goniometer is a device used to measure the range of motion (in degrees) of joints for either active or passive range. Shoulder flexion, extension, abduction adduction, internal rotation and external rotation will be assessed by Goniometer

SECONDARY OUTCOMES:
Scapular upward rotation | 4 weeks
  The Plurimeter-V gravity inclinometer will be used effectively and reliably for measuring upward rotation of the scapula in all ranges of shoulder abduction in the coronal plane
Lateral scapular slide test | 4 weeks
  The three test positions will be used. For test position one (LSST-1), the subjects were instructed to keep their upper extremities relaxed at their sides. For test position two (LSST-2), the subjects were instructed to actively place both hands on the ipsilateral hips, and consequently, the humerus was positioned in medial rotation at 45° of abduction in the coronal plane. For test position three (LSST-3), the subjects were instructed to actively extend both elbows and to elevate both upper extremities to 90° in the coronal plane with maximal internal rotation. In this procedure, the distance between inferior aspect of the inferior angle of the scapula and the closest spinous process in the same horizontal plane was measured bilaterally with a tape measure for all three positions. A difference of 1.5 cm or more in any of the three positions was considered a positive result of the LSST

CONTACTS AND LOCATIONS:
Overall Officials: Mona M ibrahim, Study Director — Cairo University; mahmoud alsehemy, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt